CLINICAL TRIAL: NCT04336618
Title: Multi-Parametric MRI Assessment of the Liver in the Dallas-FortWorth Metroplex Population
Acronym: DFWRegistry
Status: Completed | Type: Observational
Sponsor: Perspectum (Industry)
Responsible Party: Sponsor
Other Study IDs: EC-236
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Liver MultiScan — The LiverMultiscan is a quick 15 minute, contrast free, non-invasive MRI scan that provides 3 liver metrics

SUMMARY:
To build a Registry of volunteers by inviting them to get a LiverMultiScan(LMS)and collecting their contact information to seek interest in participating in future studies.

DETAILED DESCRIPTION:
This is a Registry where there will be no intervention to the standard of care.Participants will be required to attend a single visit that will involve having a multi-parametric MRI at no cost to them. In addition, the invesigators will collect contact information of participants including their email address, phone number and house address so that they can be contacted to discuss possible participation in future studies which may be sponsored by Perspectum or third parties, such as pharmaceutical companies, the participants personal information shall never be shared with these third-parties. Additionally, the contact information of the participants medical providers shall be collected so that, if requested, their LMS reports can be used in their diagnostic pathway.

Imaging will be performed at two Touchstone Imaging locations, one in downtown Dallas and the other in Southlake.

A total of 100 participants will be enrolled over a period of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers aged 18 years and over•
* Participant willing and able to give informed consent for participation in the registry.

Exclusion Criteria:

* The participant may not enter the Registry if they have any contraindication to magnetic resonance imaging (standard MR exclusion criteria at the imaging center including pregnancy, extensive tattoos, pacemaker, shrapnel injury, severe claustrophobia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult volunteers willing to get an MRI scan for the assessment of their liver
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
To build a Registry of volunteers by inviting them to get a LiverMultiScan(LMS)and collecting their contact information to seek their interest in participating in future studies | 12 months

SECONDARY OUTCOMES:
To use multi-parametric MRI (LMS) of the liver to assess the volunteer's liver health | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Perspectum Inc., Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided